CLINICAL TRIAL: NCT01568775
Title: An Open-label, Parallel Group, Single-sequence Study to Evaluate Pharmacokinetics, Safety, and Tolerability of a Single Dose Administration of Aliskiren (SPP100) in Patients With End Stage Renal Disease on Hemodialysis and Matched Healthy Subjects
Brief Title: Pharmacokinetics, Safety and Tolerability of Aliskiren (SPP100) in Patients With End Stage Renal Disease on Hemodialysis and Matched Healthy Subjects
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Novartis (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None
Other Study IDs: CSPP100A2262; 2009-014358-13 (EudraCT Number)
Record Dates: First submitted 2012-03-29; First posted 2012-04-02 (Estimated); Last update posted 2012-04-02 (Estimated); Status verified 2012-03

CONDITIONS: End Stage Renal Disease
Keywords: End Stage Renal Disease; Dialysis; aliskiren; SPP100A
MeSH Terms: conditions — Kidney Failure, Chronic | interventions — aliskiren

ARMS (1):
- Aliskiren (Experimental): All patient and subjects received single dose of aliskiren 300 mg in treatment period.
  Interventions: Drug: Aliskiren

INTERVENTIONS:
Drug: Aliskiren — All patient and subjects received single dose of aliskiren 300 mg in treatment period.
  Other Names: SPP100

SUMMARY:
This study will assess the pharmacokinetics, safety and tolerability of aliskiren in healthy subjects and patients with End Stage Renal Disease on hemodialysis.

ELIGIBILITY:
Inclusion Criteria:

1. Female subjects must be of non-child bearing potential, defined as postmenopausal women with no regular menstrual bleeding for at least 1 year prior to screening or female subjects surgically sterilized at least 6 months prior to screening. All female subjects must have negative pregnancy results at screening.
2. Subjects must weigh at least 50 kg to participate in the study, and must have a body mass index (BMI) within the range of 18 to 30 kg/m2
3. Vital signs after 3 minutes resting in the supine position (laying down) should be within the following ranges:

   * Oral body temperature between 35.0-37.8ºC
   * Systolic blood pressure, 95-140 mmHg
   * Diastolic blood pressure, 60-90 mmHg Blood pressure and pulse will be taken again in the standing position. After 3 minutes standing, there shall be no more than a 20 mm Hg drop in systolic or 10 mmHg drop in diastolic blood pressure associated with symptomatic postural hypotension.
4. Subjects must be able to communicate well with the investigator, to understand and comply with the requirements of the study. Subjects must be able to understand and sign the written informed consent.
5. Health subjects must be in good health as determined by past medical history, physical examination, vital signed assessments, electrocardiogram, and laboratory tests at screening.
6. Patients with End Stage Renal Disease who have been on intermittent hemodialysis three times a week for at least three months and are in relatively good health.

Exclusion Criteria:

1. Smokers who report cigarette use of more than 5 cigarettes per day.
2. Use of aliskiren within 2 weeks prior to study entry.
3. Participation in any clinical investigation within 3 months prior to initial dosing.
4. Hemoglobin levels outside 11-14 mg/dL
5. A history/presence of diabetes mellitus
6. A past medical history of arrhythmias, heart failure, unstable angina pectoris, stroke, or myocardial infarction within 6 months of the start of the study.
7. A past medical history of significant electrocardiogram abnormalities.
8. Recent (within the last 3 years) and/or recurrent history/presence of autonomic dysfunction (e.g., recurrent episodes of fainting, palpitations, etc).
9. Recent (within the last 3 years) and/or recurrent history/presence of acute or chronic bronchospastic disease (including asthma and chronic obstructive pulmonary disease, treated or not treated).
10. Significant drug allergy or history of atopic allergy (asthma, urticaria, eczematous dermatitis). A known hypersensitivity to aliskiren.
11. Total white blood cell (WBC) count outside the normal laboratory reference range.
12. History of immunodeficiency diseases, including a positive HIV (ELISA and Western blot) test result.
13. A positive Hepatitis B surface antigen or Hepatitis C test result.
14. History of drug or alcohol abuse within the 12 months prior to dosing, or evidence of such abuse as indicated by the laboratory assays conducted during the screening on Day -1 of each treatment period.
15. Consumption of grapefruit or grapefruit juice within 14 days prior to dosing.
16. Lactating and breastfeeding females.
17. History of head and neck angioedema.
18. Donation or loss of 400 mL or more of blood within 8 weeks prior to initial dosing.

Other protocol-defined inclusion/exclusion criteria may apply

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 12 (Actual)
Dates: Start 2010-06; Primary Completion 2010-09 (Actual); Study Completion 2010-09 (Actual)

PRIMARY OUTCOMES:
Measure: Pharmacokinetics of aliskiren: Area under the concentration-time curve from time zero to 48- hour post-dose (AUC(0-48hrs)), from time zero to the last measurable concentration sampling time (AUClast), from time zero to infinity (AUCinf) | 48 hours (period 1) , 1 hour (Period 2)
  Pharmacokinetics (concentrations of aliskiren in blood and urine) of a single dose of aliskiren in End Stage Renal Disease (ESRD) patients on hemodialysis and matched healthy subjects was analyzed.
Pharmacokinetics of aliskiren: Maximum (peak) observed blood and urine drug concentration (Cmax) after single dose administration | 48 hours (period 1) , 1 hour (Period 2)
  Pharmacokinetics (concentrations of aliskiren in blood and urine) of a single dose of aliskiren in End Stage Renal Disease (ESRD) patients on hemodialysis and matched healthy subjects was analyzed.
Pharmacokinetics of aliskiren: Time to reach maximum (peak) blood and urine drug concentration (Tmax) and elimination half-life (t1/2) after single dose administration | 48 hours (period 1) , 1 hour (Period 2)
  Pharmacokinetics (concentrations of aliskiren in blood and urine) of a single dose of aliskiren in End Stage Renal Disease (ESRD) patients on hemodialysis and matched healthy subjects was analyzed.

SECONDARY OUTCOMES:
Effect of timing of hemodialysis on the PK of aliskiren in End Stage Renal Disease (ESRD) patients | 48 hrs (Period 1), 1 hr (Period 2)
Number of patients with adverse events, serious adverse events and death | maximum 30 days

CONTACTS AND LOCATIONS:
Locations (1):
- Charité Universitätsmedizin, Berlin, Germany